CLINICAL TRIAL: NCT07194590
Title: Equol Supplementation for Improving Vascular Function in Postmenopausal Women With CKD
Brief Title: Equol and Vascular Function in Women With Chronic Kidney Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25-0095
Record Dates: First submitted 2025-09-12; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Chronic Kidney Disease (Stage 3-4); Vascular Function; Cognitive Functions; Cerebrovascular Function; Blood Pressure
Keywords: S-equol; Randomized Controlled Trial; Chronic Kidney Disease; Women's Health; Vascular Function
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Equol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Equol (Experimental): This group will receive 10 mg equol per day (2 capsules/day, 5mg equol/capsule).
  Interventions: Drug: Equol
- Placebo (Placebo Comparator): This group will receive 2 placebo capsules per day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Equol — This group will receive 10 mg equol per day (2 capsules/day, 5mg equol/capsule).
  Other Names: Equelle
  Arms: Equol
Drug: Placebo — This group will receive 2 placebo capsules per day.
  Arms: Placebo

SUMMARY:
The risk of cardiovascular disease (CVD) is significantly elevated in patients with chronic kidney disease (CKD). Notably, women with CKD commonly experience menstrual disturbances induced by CKD, which may contribute to impaired vascular function and elevated CVD risk. However, most of the literature in nephrology focuses on male patients, and studies on women's vascular health are limited. Establishing effective therapies for improving vascular function and reducing CVD risk in women with CKD is a high research priority of the NIH.

Equol contributes to improvement in vascular function, mediated in part by its anti-oxidative and anti-inflammatory properties. However, there is no information on the effect of equol on vascular function in women with CKD. The proposed project aims to determine the effect of 12 weeks of oral equol supplementation on vascular function in postmenopausal women with CKD.

DETAILED DESCRIPTION:
Patients with chronic kidney disease (CKD) have a significantly higher risk of cardiovascular diseases (CVD). Indeed, CVD is the leading cause of death in these patients. A primary reason why CKD so greatly exacerbates CVD risk is that CKD accelerates vascular dysfunction, including endothelial dysfunction (i.e., reduced brachial artery flow-mediated dilation [FMDBA]) and increased arterial stiffness (i.e., reduced compliance of the large-elastic arteries such as carotid artery), mediated in part by oxidative stress and inflammation that subsequently reduce the bioavailability of nitric oxide (NO; a vasodilator). Given CKD affects 15% of the U.S. population and 13% of the global population, CKD and its associated CVD risk are major public health concerns.

Women with CKD commonly experience menstrual disturbances, amenorrhea, and/or early menopause. Impaired ovarian function is well-known to compromise vascular health and increase CVD risk even in healthy women. As such, the vasculature of women with CKD may be exposed to the detrimental effects of both CKD and impaired ovarian function, which is secondary to CKD and menopause. Thus, declining kidney function and reduced circulating levels of cardioprotective sex hormones, particularly estradiol (E2), are two interrelated factors that contribute to vascular dysfunction and elevated CVD risk in women with CKD.

The long-term use of hormone replacement therapy (HRT) in postmenopausal women is controversial due to studies reporting its adverse effects on cardiovascular risk and breast cancer, which resulted from the long-term use of HRT. Current guidelines reserve the use of HRT only for short-term treatment of menopausal symptoms (e.g., vasomotor), prevention of bone loss and fractures, hypoestrogenism caused by hypogonadism, surgical menopause, or primary ovarian insufficiency. In women with CKD, limited studies examined the effect of HRT. Given reduced vascular dysfunction (associated with reduced circulating E2 secondary to CKD and menopause) and high CVD risk in postmenopausal women with CKD, there is a strong need for the identification of alternative pharmacological compounds to HRT that can improve vascular function in this population.

Equol is a gut microbiota-derived secondary metabolite of soy isoflavone (i.e., daidzein). Equol has been identified as a vasoactive nutraceutical and has been shown to benefit vascular function in preclinical studies and clinical studies including healthy subjects. Similar to E2, the beneficial effect of equol on vascular function appears to be in part mediated by its anti-inflammatory and anti-oxidative properties that subsequently increase NO production. However, whether equol improves vascular function in postmenopausal women with CKD is unknown.

The overall goal is to examine the efficacy and underlying mechanisms of a novel therapeutic intervention - oral supplementation with equol - for improving CKD-associated vascular dysfunction in women. In a parallel, placebo-controlled, double-blind (RCT), the longer term effects (12 weeks) of equol supplementation on vascular function will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* Aged ≥50 years
* CKD stage 3 or 4 (eGFR with the CKD-EPI 2021 race-free equation: 15-59 mL/min/1.73m2; stable renal function in the past 3 months)
* Low habitual intake of soy (soy-related food intake < 2 times per week assessed by Soy-Specific Food Frequency Questionnaire)
* Weight stable in the prior 3 months (<2 kg weight change) and willing to remain weight stable throughout the study
* Ability to provide informed consent.

Exclusion Criteria:

* Patients with advanced CKD requiring chronic dialysis
* Uncontrolled hypertension in CKD group (BP >140/90 mmHg)
* Use of any hormone replacement therapy
* Allergy and/or intolerance to soy or soy-based products
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), or total bilirubin values 2X upper limit of normal range (upper limit of normal range AST: 117 U/L; ALT: 52 U/L; total bilirubin: 1.3 mg/dL)
* History of breast cancer
* Significant co-morbid conditions with a life expectancy of < 1 year
* Current tobacco or nicotine use or history of use in the last 12 months
* History of kidney transplant
* History of severe congestive heart failure (i.e., ejection fraction <35%)
* History of hospitalization within the last month
* Immunosuppressant agents taken in the past 12 months
* Known malignancy

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2030-11-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
Brachial Artery Flow-Mediated Dilation (FMDBA) | Baseline, 12 weeksv
  Flow-mediated dilation of the brachial artery will be performed using ultrasonography and analyzed with a commercially available software package as percent change in diameter from baseline following reactive hyperemia.

SECONDARY OUTCOMES:
Carotid-Femoral Pulse Wave Velocity (CFPWV) | Baseline, 12 weeks
  A transcutaneous tonometer (Noninvasive Hemodynamics Workstation, Cardiovascular Engineering Inc.) will be positioned at the carotid and femoral arteries, and CFPWV will be calculated as the mean distance/time between the foot of the carotid and femoral arterial waveforms calculated over >30 heart cycles. Data will be expressed as m/s.
Casual blood pressure | Baseline, 12 weeks
  Casual (resting) measures of systolic blood pressure (mmHg) will be measured in triplicate over the brachial artery of the non-dominant arm after 5 minutes of quiet rest, with 1 minute of recovery between each measure, using an automated oscillometric sphygmomanometer.

OTHER OUTCOMES:
Carotid artery compliance | Baseline, 12 weeks
  Carotid compliance will be calculated using arterial blood volume and change in arterial blood pressure, which provides an index of local arterial stiffness. Unit: mm/mm Hg×10-1; there is no minimum or maximum; higher values indicate better function.
Beta-stiffness index | Baseline, 12 weeks
  Beta-stiffness index will be calculated using systolic and diastolic pressure, blood viscosity, and pulse pressure, which provides an index of local arterial stiffness. Unit: A.U.; there is no minimum or maximum; higher values indicate worse function.
24-Hour Ambulatory Systolic Blood Pressure | Baseline, 12 weeks
  Brachial artery systolic blood pressure (mmHg) will be measured automatically every 20 minutes for a 24-hour period by an ambulatory blood pressure monitor and will be averaged over the entire 24-hour period.
Endothelial Cell Protein Expression | Baseline, 12 weeks
  Endothelial cells will be obtained from peripheral veins via endovascular biopsy. Cells will be recovered by centrifugation, fixed with paraformaldehyde, and slides will be prepared and frozen. Slides will be stained for the primary antibody of interest and a complementary fluorescent secondary Alexafluor 657 antibody (Invitrogen). Slides will also be stained for the extracellular domain of vascular endothelial cadherin (Abcam) for positive identification of endothelial phenotype and DAPI for nuclear integrity. Images will be digitally captured and analyzed using Image J software (NIH). Values will be reported as ratios of subject endothelial cell protein expression to human umbilical vein endothelial cell (HUVEC) control cell protein expression. The abundance or expression of the following markers will be determined: NOX1, ERK1/2, eNOS, and phospho-eNOS (Ser1177).
Plasma equol | Baseline, 12 weeks
  Plasma equol concentrations will be quantified by the CU Anschutz Metabolomics MS Core using LC/MS.
Equol producing status | Baseline
  To assess equol producing status of the participants, a 3-day isoflavone challenge will be performed prior to intervention. The participants will consume 500 mL of a soymilk drink for 3 consecutive days. On the morning of the 4th day, urine samples from the participants will be collected, equol and daidzein will be measured. Equol producing ability will be determined by equol:daidzein ratio in the urine sample. A threshold value of log10-transformed urinary equol:daidzein ratio over -1.75 (absolute ratio =0.018) will be defined as an equol producer. TheCU Anschutz Metabolomics MS Core will measure equol and daidzein concentrations in the urine using LC/MS.
Safety (adverse events) | 2, 4, 6, 8, 10, 12 weeks
  Safety will be evaluated as the number of participants with treatment-related adverse events in each group.
Tolerability (drop-out due to adverse events) | 2, 4, 6, 8, 10, 12 weeks
  Tolerability will assessed as the rate at which enrolled subjects drop out due to adverse events.
Adherence | 2, 4, 6, 8, 10, 12 weeks
  Adherence to the intervention will be assessed by counting the number of returned capsules during check-in visits.
Middle cerebral artery cerebrovascular reactivity | Baseline, 12 weeks
  Change in mean blood flow velocity of the middle cerebral artery (ΔMFVMCA) in response to hypercapnia via transcranial doppler. MFVMCA will be determined for each condition by calculating the average MCAv over each cardiac cycle for the last minute of room air and 5% CO2 condition. ΔMFVMCA will be calculated as: hypercapnic MFVMCA - normocapnic MFVMCA.
Middle cerebral artery pulsatility index | Baseline, 12 weeks
  Pulsatility index of the middle cerbral artery via transcranial doppler.. No minimum or maximum values; higher score indicates worse function.
NIH toolbox cognitive function | Baseline, 12 weeks
  Total composite score using the NIH toolbox exam
Executive function | Baseline, 3 months
  Time to complete the trailmaking test part B

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in CKD. Data shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. data use agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, ICF
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).